CLINICAL TRIAL: NCT03148483
Title: Calcium and Vitamin D Supplementation and Periodontal Therapy for Improving Metabolic and Inflammatory Profile Among Pregnant Women: a Feasibility Trial (THE IMPROVE TRIAL)
Brief Title: Calcium-vitamin D & Periodontal Therapy for Improving Metabolic and Inflammatory Profile Among Pregnant Women
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other); Copenhagen University Hospital, Denmark (Other); Rio de Janeiro State University (Other); Instituto Fernandes Figueira (Other Government); University of Oxford (Other); Boston University (Other)
Responsible Party: Principal Investigator, Amanda Rodrigues Amorim Adegboye, Senior Lecturer, Principal Investigator, University of Westminster
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2602
Record Dates: First submitted 2016-10-27; First posted 2017-05-11 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Periodontitis; Inflammation
Keywords: Pregnancy outcome; Feasibility; Milk Fortification; Periodontitis; Pregnant women; Periodontal Therapy
MeSH Terms: conditions — Periodontitis; Inflammation

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Participant
Masking Description: This is a multi-component intervention. The participants will be blinded for the milk fortification component of the intervention only.
  Participants will receive daily sachets with similar appearance either with vitamin D and calcium (intervention) or flour (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early PT plus Fortified Milk (Experimental): early periodontal therapy (during pregnancy) plus fortified milk
  Interventions: Other: Early PT; Dietary Supplement: Fortified Milk
- Early PT plus Plain Milk (Experimental): early periodontal therapy (during pregnancy) plus plain milk
  Interventions: Other: Early PT; Dietary Supplement: Plain Milk
- Delayed PT plus Fortified Milk (Experimental): delayed periodontal therapy (after delivery) plus fortified milk
  Interventions: Other: Delayed PT; Dietary Supplement: Fortified Milk
- Delayed PT plus Plain Milk (Placebo Comparator): delayed periodontal therapy (after delivery) plus plain milk
  Interventions: Other: Delayed PT; Dietary Supplement: Plain Milk

INTERVENTIONS:
Other: Early PT — Women will receive conventional non-surgical periodontal therapy (PT), consisting of prophylactic dental polishing to remove the sticky bacterial film that forms on the teeth over time, scaling and root planing, as necessary throughout pregnancy, up to delivery
  Other Names: Early non-surgical periodontal therapy
  Arms: Early PT plus Fortified Milk; Early PT plus Plain Milk
Other: Delayed PT — Women will receive conventional non-surgical PT delayed until after delivery.
  Other Names: Delayed non-surgical periodontal therapy
  Arms: Delayed PT plus Fortified Milk; Delayed PT plus Plain Milk
Dietary Supplement: Fortified Milk — participants will be advised to take two servings of a powdered milk-based drink enriched with calcium and vitamin D daily during breakfast and afternoon snack or supper to avoid concomitant intake of the prenatal iron supplements routinely prescribed for consumption with hot main meals (e.g. lunch or dinner). Women will be advised to consume 20 g of commercially available semi-skimmed milk powder (provided by the study) and one sachet with 500 IU of vitamin D3 and 1,2 g of a calcium supplement from milk extract (300 mg of calcium) twice a day.
  Arms: Delayed PT plus Fortified Milk; Early PT plus Fortified Milk
Dietary Supplement: Plain Milk — Women will be advised to consume 20 g of commercially available semi-skimmed milk powder (provided by the study) and one sachet with flour (placebo).
  Other Names: non-fortified milk (placebo)
  Arms: Delayed PT plus Plain Milk; Early PT plus Plain Milk

SUMMARY:
The improvement of maternal and child health remains a key issue in global health. Production and improved accessibility of healthy and nutrient-rich milk-based products could potentially tackle health and nutrition inequalities in low-income countries.

This study will assess the acceptability of a multi-component intervention, including provision of calcium/vitamin-D fortified milk and periodontal therapy (PT), for improving maternal periodontal health and metabolic and inflammatory profiles. The IMPROVE trial is a feasibility randomised controlled trial (RCT) with parallel qualitative process evaluation. The target population is low-income, pregnant, Brazilian women, with periodontitis, who have not seen a dentist in the last 6 months. A series of focus group discussions and interviews with the target population will be conducted to identify key barriers and enablers to adoption and implementation of the intervention in prenatal clinics in Rio de Janeiro/Brazil. Participants will be allocated to 4 groups: 1) early PT (during pregnancy) plus fortified milk; 2) early PT plus plain milk; 3) delayed PT (after delivery) plus fortified milk; 4) delayed PT plus plain milk.

The final results will contribute to the understanding of the significance of calcium and vitamin D for short and long-term health and the occurrence of diseases, as well as to inform the current global debate on vitamin-D supplementation and fortification policy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 year;
* Up to 16 weeks' gestation;
* Having ≥ 20 teeth;
* Diagnosis of periodontitis (≥ 1 tooth with at least one of periodontal sites with ≥ 4 mm of clinical attachment loss and bleeding on probing on the same site);
* Not received regular dental treatment in the last 6 months (except from those who only visited the dentist for an emergency appointment e.g. tooth extraction);
* Cognitively and physically able to complete an interview and oral examination; and
* Willing to participate (including provision of blood samples)

Exclusion Criteria:

* Diagnosis of HIV/AIDS, psychosis, diabetes before pregnancy, thyroid disease, or disorders causing vitamin D hypersensitivity (e.g. sarcoidosis and other lymphomatous disorders);
* Diagnosis of lactose intolerance or milk allergy;
* History of renal stones or family history of renal stone and hyperparathyroidism;
* presence of extensive dental cavity and decay;
* Use of antibiotics or any immune-suppressants or medication known to affect vitamin D/calcium metabolism; and
* Consumption of ≥4 servings/day of dairy products or taking vitamin D supplements at > 400 IU/day.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility (acceptability of study design, recruitment strategy, random allocation and data collection procedures) | From baseline till 6-8 weeks' postpartum
  Feasibility will be evaluated using mixed-methods to explore intervention delivery, participants' acceptability, challenges and issues faced during the study, and recommended changes to the study design.
  Focus groups discussions will be held prior to trial recruitment to discuss issues regarding recruitment strategy, study design and data collection. In addition, group discussions will be held throughout the study (2nd and 3rd trimester) to assess potential barriers and facilitators to the intervention and data collection. At the end of each participant's involvement in the study, the participant will be asked to complete an anonymous, acceptability questionnaire to gain insights about participant's reactions to research participation and how acceptable the participant found study requirements and assessments were.
Recruitment rate | one year
  This will be measured by the total number of participants recruited into the study. The investigators intend to recruit 120 participants. Recruitment rate will be calculated (number of participants per month)
Adherence | From baseline till 6-8 weeks' postpartum
  number of drop-outs in each study arm. Analyses of drop-out rates (%) in four study arms. Self-reported quantity of milk consumed during the study. Number of follow-up visits. Proportion of participants who provide full data at baseline, throughout pregnancy and up to 6-8 weeks postpartum.

SECONDARY OUTCOMES:
Changes in % of sites with bleeding on probing | baseline and 6-8 weeks' postpartum
  Certified and calibrated dentists will conduct dental examinations pre/post-intervention. Full mouth periodontal examination will be performed at six sites per tooth, using disposable periodontal probes with coloured-coded area and mirror but without X-rays. Bleeding scores will be determined as percentage of sites with bleeding relative to the total number of sites examined.
Changes in maternal blood biomarkers to assess inflammation | 10 months on average
  Blood samples will be taken to assess changes in cytokines levels: CRP, IL-6 and MMP-9.
Changes in maternal serum levels of 25(OH)D | 10 months on average
  Blood samples will be taken to assess changes in 25(OH)D levels
Changes in maternal glucose levels | 10 months on
  Fasting blood samples will be taken to assess changes in glucose levels
Changes in maternal insulin levels | 10 months on average
  Fasting blood samples will be taken to assess changes in insulin levels
Changes in maternal serum levels of calcium | 10 months on average
  Fasting blood samples will be taken to assess changes in calcium levels
Changes in maternal blood lipids levels | 10 months on average
  Fasting blood samples will be taken to assess changes in total cholesterol and HDL-c
Neonatal levels of 25(OH)D | between 8 to 22 months
  drops of neonatal capillary blood will be collected via heel prick (200 μl) for measurement of 25(OH)D concentrations at the routine neonatal check-up
Neonatal levels of calcium | between 8 to 22 months
  drops of neonatal capillary blood will be collected via heel prick (200 μl) for measurement of calcium concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Municipal de Saúde de Duque de Caxias & Policlínica Hospital Duque de Caxias, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
External users will be bound by a data sharing agreement (in Portuguese and English) which will be available as part of the application to share data on the University website

REFERENCES:
- [Derived] Rodrigues Amorim Adegboye A, Cocate PG, Benaim C, da Veiga Soares Carvalho MC, Schlussel MM, de Castro MBT, Kac G, Heitmann BL. Recruitment of low-income pregnant women into a dietary and dental care intervention: lessons from a feasibility trial. Trials. 2020 Mar 5;21(1):244. doi: 10.1186/s13063-020-4142-5. PMID 32138765
- [Derived] Cocate PG, Kac G, Heitmann BL, Nadanovsky P, da Veiga Soares Carvalho MC, Benaim C, Schlussel MM, de Castro MBT, Alves-Santos NH, Baptista AF, Holick MF, Mokhtar RR, Bomfim AR, Adegboye ARA. Calcium and vitamin D supplementation and/or periodontal therapy in the treatment of periodontitis among Brazilian pregnant women: protocol of a feasibility randomised controlled trial (the IMPROVE trial). Pilot Feasibility Stud. 2019 Mar 5;5:38. doi: 10.1186/s40814-019-0417-6. eCollection 2019. PMID 30873290